CLINICAL TRIAL: NCT06330675
Title: Safety and Benefits of Mobilization at 4 Hours Compared to 24 Hours After Implantation of an Intracardiac Electronic Device: a Randomized Clinical Trial of Non-inferiority, Open and Controlled in Parallel Groups
Brief Title: Correct Mobilization Time After Implantation of an Intracardiac Electronic Device Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caporali Elena (Other)
Collaborators: Cardiocentro Ticino (Other)
Responsible Party: Sponsor-Investigator, Caporali Elena, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01820
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pacemaker; Defibrillators, Implantable
Keywords: Pacemaker; Implantable cardioverter-defibrillator; Early mobilization; Bed-rest
MeSH Terms: interventions — Early Ambulation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobilization 4-h after procedure (Experimental): Short-term bed-rest (4-h) after CIED implantation
  Interventions: Other: Early mobilization
- Mobilization day-after procedure (Active Comparator): Standard of care with prolungate bed-rest after CIED implantation
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Early mobilization — Short-term bed-rest and immobilization
  Arms: Mobilization 4-h after procedure
Other: Standard of care — Bed-rest and immobility until the day-after procedure
  Arms: Mobilization day-after procedure

SUMMARY:
Bedrest is usually prescribed for patients management after cardiac electronic device implantation (CIED) in order to prevent complication. Due to the lack of guidelines available on the timing of postoperative mobilization management, the aim of the study is to evaluate the safety of early mobilization, comparing mobilization at 4-h against day-after procedure.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Signed informed consent form
* New permanent pacemaker implantation (PM) or implantable cardioverter-defibrillator (ICD)

Exclusion Criteria:

* CIED implants after recent cardiac surgery
* Upgrade or revision of implanted device
* CRT implantation
* Intraoperative complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint: pacing lead dislodgement, pocket hematoma, pneumothorax, and pericardial effusion | Within 48 hours post operative
  Incidence of post-operatory complications (composite endpoint). Non inferiority margin 5%

SECONDARY OUTCOMES:
Post-operative pain | 24 hours
  Pain will be assessed with the Numerical Rating Scale (NRS) scale ranging from 0 to 10 (0 corresponds to no pain and 10 to maximal level of pain).
Sleep disturbance | The first night after surgery
  Quality of sleep will be assessed using the Richards-Campbell Sleep Questionnaire (RCSQ), which ranges from 0 to 500 points, where 0 indicates the worst possible sleep quality and 500 the best possible. The sub-scores include sleep depth, sleep latency, number of awakenings, return to sleep after awakening, and overall sleep quality (each ranging from 0 to 100 points).
Number of participants with postoperative urinary retention | Within 24 hours post operative
  Number of participants requiring an intervention such as a Foley catheter or catheterization
Number of participants developing postoperative delirium | Within 24 hours post operative
  Number of participants who develop postoperative delirium, as assessed by the 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM)
Number of participants developing orthostatic intolerance | First out-of-bed mobilization
  Number of participants who develop symptoms of orthostatic intolerance such as dizziness, nausea, vomiting, blurred vision, or syncope, during mobilization
Quality of recovery | Day 1
  Quality of recovery assessed with the Quality of recovery-15 (QoR-15) ranging from 0 (extremely poor quality of recovery) to 150 (excellent quality of recovery), and sub-scores (physical comfort 0-50, emotional state 0-40, psychological support 0-20, physical independence 0-20 and pain 0-20).
Number of participants developing pressure ulcer | Within 48 hours post operative
  Number of participants who develop pressure ulcers, assessed using Pressure Ulcer Classification System (stage 1, stage 2, stage 3, and stage 4)

OTHER OUTCOMES:
Incidence of pacing lead dislodgement, pocket hematoma, pneumothorax, pericardial effusion, and pocket infection | 3 month
  Number of patients suffering with post-operatory complications

CONTACTS AND LOCATIONS:
Overall Officials: Elena Caporali, MD, Principal Investigator — Cardiocentro Ticino Institute - EOC
Locations (1):
- Cardiocentro Ticino Institute - EOC, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No